CLINICAL TRIAL: NCT07318051
Title: Sample Collection for Ongoing Research and Product Evaluation (SCORE) Study
Brief Title: Sample Collection for Ongoing Research and Product Evaluation Study
Acronym: SCORE
Status: Recruiting | Type: Observational
Sponsor: Natera, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 25-081-NCP
Record Dates: First submitted 2025-12-19; First posted 2026-01-05 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer; Lung Cancer; Muscle Invasive Bladder Cancer; Rectal Cancer; Pancreatic Cancer; Ovarian Cancer; Gastroesophageal Cancer; Prostate Cancer; Melanoma; Head and Neck Cancer; Uterine Cancer; Liver Cancer
Keywords: Breast cancer; Lung cancer; Muscle invasive bladder cancer; Rectal cancer; Pancreatic cancer; Ovarian cancer; Gastroesophageal cancer; Prostate cancer; Melanoma; Head and Neck cancer; Uterine cancer; Liver cancer
MeSH Terms: conditions — Breast Neoplasms; Lung Neoplasms; Rectal Neoplasms; Pancreatic Neoplasms; Ovarian Neoplasms; Prostatic Neoplasms; Melanoma; Head and Neck Neoplasms; Uterine Neoplasms; Liver Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood and tissue samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The SCORE study is a prospective, multi-site clinical trial designed to collect blood and tissue samples, along with relevant clinical data, from participants diagnosed with various solid tumors. The collected specimens and information will be used to evaluate the clinical performance of Natera's molecular residual disease (MRD) testing across multiple cancer types. The study aims to assess the ability of Natera's assays to detect circulating tumor DNA (ctDNA) as a marker for disease recurrence and treatment response.

DETAILED DESCRIPTION:
The study is designed to evaluate the clinical performance of Natera's molecular residual disease (MRD) assays in detecting ctDNA across multiple solid tumor types. The goal is to assess the ability of the assay to identify minimal residual disease, monitor disease recurrence, and evaluate treatment response following standard-of-care therapy. No individual test results from the study testing will be provided to participants or their treating clinicians.

Participants who meet eligibility criteria for the SCORE study will be invited to enroll and must provide written informed consent prior to undergoing any study procedures. Participants will provide study-specific blood samples.

The SCORE study includes three participant cohorts:

* Cohort A - Surgical with Curative Intent
* Cohort B - Neoadjuvant Therapy
* Cohort C - Metastatic/No Surgery

Participants may be followed for up to eight years. During the first three years, blood samples will be collected periodically, approximately every six weeks, for up to two years after surgery or completion of primary treatment. Participants will have data-only follow-up visits at one and five years after the final blood collection.

Tissue Sample Collection Residual tissue samples, collected as part of standard-of-care procedures, will also be obtained for study purposes.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older.
2. Any patient that has an untreated primary solid malignancy within the following cohorts:

   1. Breast cancer
   2. Lung cancer
   3. Muscle invasive bladder cancer
   4. Rectal cancer
   5. Pancreatic cancer
   6. Ovarian cancer
   7. Gastroesophageal cancer
   8. Prostate cancer
   9. Melanoma
   10. Hepatic/liver cancer
   11. Uterine/endometrial cancer
   12. Head and neck Cancer
3. The participant has a suspected primary malignancy of pancreatic, endometrial, bladder, or ovarian cancer based on imaging.
4. Eastern Cooperative Oncology Group performance status ≤ 2.
5. Able to tolerate venipuncture for research blood draw(s).
6. Consent to provide residual tumor tissue for research.
7. Willing and able to comply with the study requirements.
8. Signed informed consent(s) must be obtained prior to participation in the study.

Exclusion Criteria:

1. Pregnant or breastfeeding.
2. Prior history and treatment for any cancer within the past year or has another active cancer, with the exception of participants who have undergone surgical removal of skin squamous cell or basal cell cancers.
3. Has initiated postoperative systemic treatment.
4. At time of enrollment, has undergone or plans to undergo any ctDNA testing to assess molecular residual disease, with the exception of comprehensive genomic profiling for therapeutic selection.
5. History of bone marrow or organ transplant.
6. Serious medical conditions that may adversely affect ability to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants 18 years of age or older diagnosed with malignant, invasive solid tumors prior to receiving treatment.
Sampling Method: Non-Probability Sample
Enrollment: 9600 (Estimated)
Dates: Start 2025-07-21 (Actual); Primary Completion 2035-01 (Estimated); Study Completion 2035-01 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome - Collection of Blood and Residual Tissue Specimens for Cancer Assay Development | 8 years
  To collect de-identified whole blood and residual tissue specimens for research use and the development of blood-based cancer monitoring and detection assays.

SECONDARY OUTCOMES:
Secondary Outcome - Collection of Blood and Residual Tissue Specimens for Disease Assay Development | 8 years
  To collect de-identified whole blood and residual tissue specimens for research use and the development of blood-based disease assays.

CONTACTS AND LOCATIONS:
Locations (1):
- Natera, Inc., Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No